CLINICAL TRIAL: NCT02489994
Title: Clinical Study to Evaluate the Performance of the ePrime System for the Treatment of Cellulite
Brief Title: Performance of the ePrime System for Cellulite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF15911
Record Dates: First submitted 2015-06-25; First posted 2015-07-03 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all subjects (Experimental): Treatment with the ePrime radiofrequency microneedling device in the upper thighs and buttocks
  Interventions: Device: ePrime

INTERVENTIONS:
Device: ePrime — The main intent of the ePrime for cellulite is to utilize a minimally-invasive approach to directly deliver RF energy into tissue through pairs of micro-electrode needles and use temperature sensors within the needles to reliably create fractional thermal injuries within the skin.

SUMMARY:
Clinical Study to Evaluate the Performance of the ePrime System for the Treatment of Cellulite.

DETAILED DESCRIPTION:
Up to 60 healthy adult volunteers seeking cellulite treatment, females of 25 to 60 years of age, from multiple investigational sites.

This is an open-label, multi-center study. Subjects in this study will receive a single subcutaneous treatment with the ePrime device in one treatment session according to the study protocol.

Prior to treatments, tissue to be treated will be injected with tumescence or local dermal infiltration solution according to the protocol. Subjects will return for follow-up (FU) visits at: 1 week, 1 month, 3 months and 6 months following the treatment.

Methodology described in protocol to evaluate efficacy of treatments will be carried out at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects seeking treatment of cellulite in the upper thighs and buttocks areas.
2. Subject have cellulite stage II or III as graded using Nurnberger-Muller scale clasification (Appendix III)
3. Healthy female subjects ages 25 to 60 years of age
4. Informed consent process completed and subject signed consent
5. Willing to receive the proposed ePrime treatment and follow-up protocol
6. Not pregnant or lactating and must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence)
7. Willing to have photographs taken of the treated areas to be used de-identified in evaluations, publications and presentations

Exclusion Criteria:

1. Subject had surgery or any other procedure for cellulite in the last 6 months
2. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding
3. Known allergy to lidocaine or epinephrine or antibiotics
4. Active malignancy or history of malignancy in the past 5 years
5. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator
6. Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), lupus, porphyria, or pertinent neurological disorders (i.e. any disease state that in the opinion of the Physician would interfere with the anesthesia, treatment, or healing process)
7. Having a known anticoagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of use as per the subject's physician discretion)
8. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications
9. Suffering from hormonal imbalance, whether related to thyroid, pituitary, or androgen
10. History of significant lymphatic drainage problems
11. History of cancer which required lymph node biopsy or dissection
12. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions, hidradenitis, or dermatitis of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
13. History of keloid scarring, abnormal wound healing and / or prone to bruising
14. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders
15. Use of isotretinoin (Accutane®) within 6 months of treatment or during the study
16. Subject on systemic corticosteroid therapy 6 months prior to and throughout the course of the study
17. Dysplastic nevi in the area to be treated
18. Participation in a study of another device or drug within 3 month prior to enrollment or during this study, if treatments of cellulite were involved
19. Subject has palpable lymphadenopathy at any visit. Standard palpation techniques will be used
20. Subjects with history of severe edema
21. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2014-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Improvement in cellulite compared to baseline for the upper thighs and buttocks, as assessed by blinded evaluation of clinical photographs | Baseline and 3 months post treatment visit
  Evaluate the efficacy of a single dermal and subcutaneous treatment with ePrime for the upper thighs and buttocks cellulite as assessed by blinded evaluators at 3 months post treatment visit.

SECONDARY OUTCOMES:
Improvement in cellulite compared to baseline for the upper thighs and buttocks, as assessed by blinded evaluation of clinical photographs | Baseline and 6 months post treatment visit
  Evaluate the efficacy of a single dermal and subcutaneous treatment with ePrime for the upper thighs and buttocks cellulite as assessed by blinded evaluators at 6 months post treatment visit.
Number of Participants with Adverse Events | day 0 up to 7 months
  evaluate the safety of a single dermal and subcutaneous treatment with ePrime for the upper thighs and buttocks cellulite at 1 week post treatment, 1 month, 3 and 6 months following the treatment.
Improvement in cellulite compared to baseline | Baseline, 1 month, 3 and 6 months post treatment visit.
  Improvement in cellulite compared to baseline, as assessed by study investigators, using Nurnberger-Muller scale at 1 month, 3 and 6 months post treatment visit.
Investigator satisfaction - by questionnaire | 1, 3, and 6 months post-treatment visit
  Evaluate Investigator satisfaction at 1, 3, and 6 months post-treatment visit, using a satisfaction scale
Subject satisfaction - by questionnaire | 1, 3, and 6 months post-treatment visit
  Evaluate subject satisfaction at 1, 3, and 6 months post-treatment visit, using a satisfaction scale

CONTACTS AND LOCATIONS:
Overall Officials: Macrene Alexiades, MD, Principal Investigator — Dermatology and Laser Surgery Center 955 Park Avenue, New York, NY, 10028; Leyda Bowes, MD, Principal Investigator — Bowes Dermatology, 3659 South Miami Avenue, Suite # 6008, Miami, FL 33133; David Goldberg, MD, Principal Investigator — Skin Laser & Surgery Specialist of NY/NJ; Girish Munavalli, MD, Principal Investigator — Laser & Vein Specialists of the Carolinas, 1918 Randolph Road, Suite 550, Charlotte, NC 28270
Locations (4):
- United States (4):
  - Bowes Leyda, Miami, Florida
  - David Goldberg, Hackensack, New Jersey
  - Macrene Alexiades, New York, New York
  - Girish Munavalli, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rawlings AV. Cellulite and its treatment. Int J Cosmet Sci. 2006 Jun;28(3):175-90. doi: 10.1111/j.1467-2494.2006.00318.x. PMID 18489274
- [Background] Rossi AB, Vergnanini AL. Cellulite: a review. J Eur Acad Dermatol Venereol. 2000 Jul;14(4):251-62. doi: 10.1046/j.1468-3083.2000.00016.x. PMID 11204512